CLINICAL TRIAL: NCT06514313
Title: Phase II Randomized Controlled Clinical Trial of Mitoxantrone Hydrochloride Liposome Combined With Irinotecan and Vincristine (VIM) With VIT in Children With Relapsed and Refractory Soft Tissue Sarcoma.
Brief Title: Clinical Trial of VIM With VIT in Children With Relapsed and Refractory Soft Tissue Sarcoma.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yizhuo Zhang (Other)
Responsible Party: Sponsor-Investigator, Yizhuo Zhang, Director, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-STS-K01
Record Dates: First submitted 2024-07-04; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIM (Experimental): Mitoxantrone Hydrochloride Liposome combined with Irinotecan and Vincristine.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome+Irinotecan+Vincristine
- VIT (Active Comparator): Temozolomide combined with Irinotecan and Vincristine.
  Interventions: Drug: Temozolomide+Irinotecan+Vincristine

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome+Irinotecan+Vincristine — Mitoxantrone hydrochloride liposome will be administered by an intravenous infusion , 4 cycles.
  Arms: VIM
Drug: Temozolomide+Irinotecan+Vincristine — Q3W, 4 cycles
  Arms: VIT

SUMMARY:
Explore the efficacy and safety of mitoxantrone liposome combined with irinotecan and vincristine (VIM) in the treatment of relapsed/refractory soft tissue sarcoma in children.

DETAILED DESCRIPTION:
Children with relapsed/refractory soft tissue sarcoma who meet the inclusion criteria are randomly divided into VIM group and VIT group (irinotecan, vincristine, temozolomide) at 1:1. The efficacy and safety of the two groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* 2 years ≤age≤21 years, no gender limitation.
* The Karnofsky (≥16 years old) or Lansky (< 16 years old) physical status score is at least 70.
* The expected survival time is not less than 12 weeks.
* Heart function: a) Cardiac COLOR ultrasound detection LVEF≥ 50%; b) ECG suggests no myocardial ischemia; c) No history of arrhythmia requiring drug intervention before enrollment.
* Pathological results for patients of soft tissue sarcoma.
* Patients with rhabdomyosarcoma are limited to first -, second -, and third-line treatment, and patients with other pathological subtypes are limited to progression, recurrence, or refractory after first-line treatment, with refractory defined as failure to achieve complete or partial response to the most recent treatment.
* Measurable lesions (according to RECIST 1.1 standards, measurable lesions have not received radiotherapy, freezing and other local treatments).
* The patient must fully recover from the acute toxic effects of all previous anticancer chemotherapy.
* Good blood and organ function.
* During study participation, patients are able to adhere to outpatient treatment, laboratory monitoring, and necessary clinical visits.
* The parent/guardian of the child or adolescent subject is capable of understanding, agreeing to, and signing the study Informed consent (ICF) and the applicable child consent form prior to initiating any program-related procedures; Subject is capable of expressing consent with parental/guardian consent (if applicable).

Exclusion Criteria:

* Once received mitoxantrone or mitoxantrone liposomes.
* Patients who had received previous VIT (irinotecan + temozolomide + vincristine) chemotherapy.
* Previous treatment with adriamycin or other anthracyclines with a total cumulative dose of adriamycin > 360 mg/m^2; Or patients with cardiac disease caused by previous anthracyclines.
* Receiving or not being able to discontinue P450 enzyme-induced anticonvulsant drugs (e.g., phenytoin, carbamazepine, etc.) within 4 weeks or 5 half-life periods prior to enrollment.
* Previous or concurrent clinical significance of active cardiovascular diseases.
* Severe chronic skin diseases in the past.
* Previous allergic asthma or severe allergic disease.
* Uncontrolled hypertension and diabetes.
* Have a history of other tumors, except cured cervical cancer or basal cell carcinoma of the skin.
* Active hepatitis B or hepatitis C infection.
* HIV or syphilis infected patients.
* Patients who have previously received organ transplants.
* Uncontrolled active systemic bacterial, viral, or fungal infection.
* Contraindications to high-dose hormone use, such as uncontrolled hyperglycemia, gastric ulcers, or psychiatric disorders.
* Severe neurological or psychiatric history, including epilepsy or autism.
* Pregnant, lactating women and patients of childbearing age who are unwilling to use contraception.
* Other circumstances deemed inappropriate by the investigator to participate in the study.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 cycles of chemotherapy (each cycle is 21 days)
  Objective response rate (ORR) after 2 cycles of chemotherapy with VIM or VIT regimen, including complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 4 cycles of chemotherapy (each cycle is 21 days)
  Objective response rate (ORR) after 4 cycles of chemotherapy with VIM or VIT regimen, including complete response (CR) and partial response (PR)
Disease control rate (DCR) | Up to 4 cycles of chemotherapy (each cycle is 21 days)
  Refers to the percentage of patients with confirmed complete response, partial response, and disease stability in patients with evaluable efficacy
Progression-free survival (PFS) | From date of radomization unit the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 moths.
  Means from the date of enrollment to the date of first disease progression or death from any cause, whichever comes first. If the subject has no disease progression during the trial period, PFS is defined as the last date until the subject's last confirmed progression-free survival.
Overall survival (OS) | From date of radomization unit the date of first documented date of death from any cause, assessed up to 24 moths
  Overall survival (OS) was defined from the date of enrollment to the date of death from any cause.

OTHER OUTCOMES:
Circulating tumor DNA (ctDNA) . | Assessed up to 24 moths.
  ctDNA was dynamically monitored and the correlation between ctDNA and efficacy was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No